CLINICAL TRIAL: NCT05505851
Title: Sequential Core Stability Corrective Exercise Approach for Alignment And Muscle Function In Lower Crossed Syndrome
Brief Title: Sequential Core Stability Corrective Exercise Approach in Lower Crossed Syndrome
Acronym: SCSCRLCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/1104
Record Dates: First submitted 2022-05-23; First posted 2022-08-18 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Low Back Pain
Keywords: Alignment; Core Stability; Diaphragm; Pelvic floor; Dysfunction
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: 2
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: Control (Active Comparator): Corrective Exercises:
  Hip Flexor Stretch, Thoracolumbar Extensor Stretch, Abdominal Curl, and Glute Bridge.
  Interventions: Other: Control
- B: Sequential Core Stability Corrective Exercise Approach (Experimental): Sequential Core Stability Corrective Exercise Approach
  1. Corrective Exercises
  2. Diaphragm Training Program
  3. Pelvic floor Muscle training
  4. Core Stability exercises
  Interventions: Other: Sequential Core Stability Corrective Exercise Approach

INTERVENTIONS:
Other: Control — Corrective Exercises: Hip Flexor Stretch, Thoracolumbar Extensor Stretch, Abdominal Curl, and Glute Bridge.
  Arms: A: Control
Other: Sequential Core Stability Corrective Exercise Approach — Sequential Core Stability Corrective Exercise Approach
  1. Corrective Exercises
  2. Diaphragm Training Program
  3. Pelvic floor Muscle training
  4. Core Stability exercises
     1. Beginning
     2. Progressing
     3. Advanced
  Arms: B: Sequential Core Stability Corrective Exercise Approach

SUMMARY:
The objective of the study will be to determine the effects of Sequential Core Stability Corrective Exercise Approach for Alignment and Muscle Function in Lower Crossed Syndrome.

DETAILED DESCRIPTION:
Lower Crossed Syndrome is one of common postural disorder which occurs due to the muscular imbalance. It refers to specific altered muscle activation and movement patterns along with some postural deviations. Alterations in muscle activation include overactivity of hip flexors and lower back muscles paired underactivity of abdominals and gluteus muscle. This pattern of imbalance creates dysfunction. Postural correction exercise with inner and outer core muscles are necessary. There are different traditional structural approach, functional approach and biomechanics and are presumed to lead to adjustments in the length and strength of local muscles while ignoring other related malalignments and core stability. The objective of the study will be to determine the effects of Sequential Core Stability Corrective Exercise Approach for Alignment and Muscle Function in Lower Crossed Syndrome.

It will be a randomized controlled trial. Sample size will be collected after running the pilot study. The participants will be recruited through convenient sampling technique and then allocated randomly to Groups. Outcome measures will be alignment and muscle function. Pre and post reading and after one month follow-up will be recorded. Data will be analyzed using statistical package for social sciences software version 25. After assessing normality of data by Shapiro-Wilk test, it will be decided either parametric or nonparametric test will be use within a group or between two groups.

Keywords: Alignment, Core Stability, Diaphragm, Muscular Imbalance, Muscle thickness Pelvic floor.

ELIGIBILITY:
Inclusion Criteria:

* • Age group between 18 to 28 years

  * No current incidence of low back pain or past history of low back dysfunction
  * Kendall double leg lowering test: Abdominal muscle weakness to the extent of not being able to maintain posterior pelvic tilt during a double leg lowering test in supine position.
  * Diagnosed with lower cross syndrome through assessment criteria of Janda muscle testing and assessment

Exclusion Criteria:

* • Having any history of low back pain, spinal trauma,

  * Joint dysfunction in past 3 months
  * Congenital deformities at hip or lumbar region,
  * Recent fracture to related joints in past 6 months
  * Any family history of cardiopulmonary disease
  * Any disease or urogenital tract
  * Participants having BMI above 30.
  * Recent history of hepatitis or Fatty liver or
  * Any athlete having high physical activity.
  * History of abdominal, hip or lumbar surgeries in past 3 months

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-02-10 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Photometry for Pelvic Tilt | Pre (0th week), Post (6th week), (12th week) Follow-up
  Angle of Pelvic tilt will be measured Through a Reliable and validated camera.
Photometry for Chest Expansion | Pre (0th week), Post (6th week), (12th week) Follow-up
  Angle of Chest expansion will be measured at Nipple line, Xiphoid level and at waist level, Through a Reliable and validated camera.
Photometry for Cervicothoracic level | Pre (0th week), Post (6th week), (12th week) Follow-up
  Angle of C7-T1 will be measured Through a Reliable and validated camera.
Photometry for Lumber flexion | Pre (0th week), Post (6th week), (12th week) Follow-up
  Angle of Lumber curve will be measured Through a Reliable and validated camera.
Diaphragmatic excursion | Pre (0th week), Post (6th week), (12th week) Follow-up
  To assess the diaphragmatic motion by M-mode US a 2.5-5 megahertz (MHz) phase array will be used.
Levator ani Excursion | Pre (0th week), Post (6th week), (12th week) Follow-up
  To assess the pelvic floor motion by M-mode US a 2.5-5 megahertz (MHz) array will be used.
Diaphragmatic thickness and thickening | Pre (0th week), Post (6th week), (12th week) Follow-up
  diaphragmatic thicknesses and thickening will be assessed by B-mode ultrasonography during various respiratory maneuvers
Levator ani thickness and thickening | Pre (0th week), Post (6th week), (12th week) Follow-up
  Levator ani thicknesses and thickening will be assessed by B-mode ultrasonography during various respiratory maneuvers
Core stability | Pre (0th week), Post (6th week), (12th week) Follow-up
  It will be measured by Pressure biofeedback unit for the transverse abdomens.

SECONDARY OUTCOMES:
Forced Vital Capacity (FVC) | Pre (0th week), Post (6th week), (12th week) Follow-up
  Pulmonary function test through spirometer, It will be measured by digital spirometer.
Forced Expiratory Volume per second FEV1 | Pre (0th week), Post (6th week), (12th week) Follow-up
  Pulmonary function test through spirometer, It will be measured by digital spirometer.
Ratio of FEV1/ FVC | Pre (0th week), Post (6th week), (12th week) Follow-up
  Pulmonary function test through spirometer, It will be measured by digital spirometer.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, PhD, Study Chair — Riphah International University; Wajeeha Zia, PhD*, Principal Investigator — Riphah International University , QIE, Campus
Locations (1):
- Al-khumeini Trust Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No